CLINICAL TRIAL: NCT07014826
Title: Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase III Clinical Trial, to Evaluate the Efficacy and Safety of HRS-5965 Capsule in Primary IgA Nephropathy
Brief Title: A Trial of HRS-5965 Capsule in Primary IgA Nephropathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5965-305
Record Dates: First submitted 2025-05-22; First posted 2025-06-11 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): HRS-5965
  Interventions: Drug: HRS-5965
- Treatment group B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-5965 — HRS-5965
  Arms: Treatment group A
Drug: Placebo — Placebo
  Arms: Treatment group B

SUMMARY:
This multicenter, randomized, double-blind, parallel, placebo-controlled study is being conducted to evaluate the efficacy, and safety of HRS-5965 capsule for primary IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent；
2. Weight ≥35 kg, Body mass index (BMI) < 37.5kg /m2;
3. Primary IgA nephropathy was confirmed by renal biopsy within 8 years;
4. 24-UPE≥ 1.0g /24h, or 24-UPCR≥ 0.8g/g at screen, and 24-UPCR≥ 0.8g/g prior to randomization;
5. eGFR≥30 ml/min/1.73m2 at screening and prior to randomization; (CKD-EPI formula)
6. A fertile female subject or a male subject whose partner is a fertile female, who has not had a fertility, sperm/egg donation plan from the signing of the informed consent to 1 month after the last dose, and voluntarily takes effective contraceptive measures (including the partner);
7. Understand the research procedures and methods, voluntarily participate in this trial, and sign the informed consent form in person.
8. Receiving optimal supportive therapy including RAS blockers and stabilizing the dose for at least 12 weeks after reaching the maximum recommended dose or the maximum tolerated dose prior to randomization;

Exclusion Criteria:

1. Allergic to any RAS blockers, investigational products, or components as evaluated by the investigator;
2. Patients with secondary IgA nephropathy as determined by the investigator;
3. IgA nephropathy with rapid decline of renal function; Kidney pathology indicated that more than 50% of the glomerulus had large crescent body formation, which may affect the study results; Tubule atrophy - interstitial fibrosis of more than 50%;
4. Patients with a history of immunodeficiency disease; Or in combination with other systemic diseases likely to cause proteinuria; Or with Nephrotic Syndrome;
5. Have any organ transplant;
6. Patients with active infection of tuberculosis within 1 year prior to screening, such as liver abscess and pyelonephritis; Or subjects with active infection who requiring intravenous antibiotic therapy within 2 weeks prior to randomization;
7. Patients with a history of malignant neoplasms;
8. Patients with a history of severe trauma or major surgery within 12 weeks prior to screening, or who plan to undergo surgery during the study period;
9. Patients with a history of blood donation or a history of severe blood loss (≥400 mL blood loss) within 12 weeks prior to screening, or who have received blood transfusions within 12 weeks prior to screening;
10. The presence of a disease or medical condition determined by the investigator might affect drug absorption, distribution, metabolism, and excretion;
11. As determined by the investigator, the subject has any of the following: progression or recovery of a disease;
12. Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), or total bilirubin exceeding 3 times the upper limit of normal (ULN) at screening;
13. Participants who have participated in a clinical trial of any drug or medical device within 12 weeks prior to randomization and are expected to have residual effects of the investigational treatment (as determined by the investigator), or who were within the follow-up period of a clinical study, or within 5 half-lives of the investigational drug, or within 30 days (whichever is older) before screening;
14. Women who are pregnant or breastfeeding;
15. A history of drug abuse;
16. Participants who received systemic glucocorticoid or immune suppressants within 12 weeks prior to randomization and are expected to have during research；
17. Participants who received biologics or cytokine inhibitor within 6 months prior to randomization and are expected to have during research；
18. Any physical or mental illness or condition that, as determined by the investigator, is likely to increase the risk of the study, affect the subject's adherence to the protocol, or prevent the subject from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Ratio of 24-hour Urinary protein to creatinine ratio (UPCR) to baseline | Baseline and Week 36
The total annualized slope of estimated glomerular filtration rate（eGFR） | Baseline and Week 104

SECONDARY OUTCOMES:
The total annualized slope of estimated glomerular filtration rate（eGFR） | up to Week 36
Proportion of subjects with 24-hour urinary protein excretion (24-UPE) < 0.5 g/d and < 0.3 g/d | up to Week 36 and Week104
Proportion of subjects with 24-UPCR declined >50% to baseline | up to Week 36 and Week104
Ratio of 24-hour Urinary protein to creatinine ratio (24-UPCR) to baseline | up to Week 36 and Week104
Ratio of 24-hour Urinary protein to Albumin Creatinine ratio (24-UACR) to baseline | up to Week 36 and Week104
Ratio of 24-hour Urinary protein excretion（24-UPE） to baseline | up to Week 36 and Week104
Change from baseline of eGFR | up to Week 36 and Week104
Change from baseline of serum creatinine | up to Week 36 and Week104

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided